CLINICAL TRIAL: NCT02763475
Title: NK Cells Infusion as Consolidation Treatment of Acute Myeloid Leukemia in Children and Adolescents
Brief Title: NK Cells as Consolidation Therapy of Acute Myeloid Leukemia in Children/Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other); Fundación Mutua Madrileña (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NKCell_LMA_2015; 2015-001901-15 (EudraCT Number)
Record Dates: First submitted 2016-04-04; First posted 2016-05-05 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia; Leukemia; Myeloid Leukemia
Keywords: Killer Cells, Natural; Consolidation treatment; cytologic remission; Haploidentical NK Cells; allogeneic; IL-2 Expanded NK Cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Leukemia, Myeloid | interventions — Cyclophosphamide; fludarabine; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Natural Killer (NK) Cells + Chemotherapy (Experimental): Starting on day -6, 60mg/Kg cyclophosphamide by vein will be administrated. Day -5 to -1 fludarabine administrated by vein at 25 mg/m2. 24-48 hours after chemotherapy completion, NK cell infusion will be injected (day 0). On day 7 a second NK cell infusion will be administrated. First infusion consist of 5x10^7/kg NK CD3-CD56+ NK cells. The second NK cell infusion will include up to 5x10^8 CD3-CD56+ cells if no treatment related toxicity occurred. Subcutaneous IL-2 (1x10^6 UI/m2) three times a week for two weeks will be administrated after first NK infusion.
  Interventions: Drug: cyclophosphamide; Drug: Fludarabine; Procedure: NK cell infusion; Drug: IL-2

INTERVENTIONS:
Drug: cyclophosphamide — 60mg/kg by vein on day -6
Drug: Fludarabine — 25mg/m2 iv daily on day -5 to -1
Procedure: NK cell infusion — * First allogeneic haploidentical NK cell iv. infusion: 5x10e7/kg, NK CD3-CD56+ immunophenotype, 24-48h after chemotherapy
  * Second allogeneic haploidentical NK cell iv. infusion: up to 5x10e8/kg, NK CD3-CD56+immunophenotype, 7 days after the first infusion.
Drug: IL-2 — 1x10^6 UI/m2 three times a week for two weeks from first NK infusion (day 0)
  Other Names: Proleukin

SUMMARY:
The main goal of this study is to evaluate the anti-relapse prophylactic activity of inoculating Natural Killer (NK) cells as consolidation therapy of acute myeloid leukemia in paediatric patients with cytologic remission. The patients included have intermediate risk of relapse and no indication for allogeneic hematopoietic stem cell transplantation.

After the standard induction and consolidation chemotherapy treatment, patients will receive five days of fludarabine to try to kill any minimal residual disease and prevent NK cell rejection. Two different NK cells infusions will be performed within one week (day 0 and 7). Interleukin 2 (IL-2) will be administrated to increase the cytotoxic activity of NK cells.

DETAILED DESCRIPTION:
Hypothesis:

NK cells are the natural defence against cancer cells. Thus, supplementing compatible NK cells from a related donor might increase the probability to eliminate any residual chemotherapy resistant cell in Acute myelogenous leukemia patients.

Description:

NK cells will be donated from a compatible family member who has a certain genetic code in their blood, called HLA, which partly matches patient genetic code, reducing any potential rejection. Interleukin-2 is co administrated during NK cell treatment to improve effectiveness.

Methodology:

The day that patient receive first NK cell infusion is called day 0. The days before are called minus days (-D). Conversely, the days after NK cell infusion are called plus days (+D).

Study administration

* After standard chemotherapy treatment against acute myeloid leukemia (AML) and restoration of haematologic normal levels, patients will receive a 60mg/kg of cyclophosphamide (day -6) and five daily intravenous cycles 25 mg/m2 of the chemotherapic fludarabine every day (day -5, -4, -3, -2, -1).
* Day 0 will be settled from 24h to 48h after fludarabine treatment completion. NK cells will be intravenous administered twice (day 0 and day 7). The first dose of NK cells (day 0) will contain up to 5x10^7 cells/kg with immunophenotype NK (CD3-CD56+). The second dose might be higher (up to 5x10^8 cells/kg) in case of no treatment related toxicity after first NK injection. In any case, no more than 1x10^6 cells/kg with an immunophenotype T (CD56-CD3+) will be administrated.
* From day 0, IL-2 1x10^6 UI/m2 subcutaneous will be administrated three times a week during two weeks.

Study visits

Before and after the treatment a bone marrow aspirate will be analyzed in order to evaluate minimal residue disease (cytology, cytometry and/or molecular studies) at least one month after NK injection. objective response rate will be reevaluated at least once a year.

Before treatment starts:

* Birthday, gender and personal medical history will be recorded
* physical examination, including measurement of the vital signs (temperature, heart and breathing rate, etc…)
* Blood and urine test
* Bone marrow aspirate in order to evaluate the basal disease

On every visit

* Physical examination and vital signs will be recorded
* Adverse event form
* Other concomitant drugs

After NK treatment

* It will be 11 visits on days +30, +60, +90, +180, +270, +360, +480, +600, +720, +900, +1080 which included a blood and urine test and Lansky/karnofsky scale.
* Additionally on days +30, +360, +720 and +1080 a bone marrow aspirate will be performed to evaluate relapse.

Length of the study:

Up to 35 AML patients will be included in the study during a 32 months recruitment period with a patient follow-up of thirty-six months. The maximum length of the study will be six years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 0 and 21 years, diagnosed with AML in first cytological remission who have completed the induction and consolidation chemotherapy phases and no criteria for allogeneic hematopoietic stem cell transplantation (HSCT), ie patients who have responded well to induction lacking donor HLA identical relative and do not have high-risk cytogenetic abnormalities.
2. Karnofsky or Lansky Performance Scale (PS) > 60%
3. Mild-moderate (<4) organ functional impairment (liver, kidney, respiratory) according to the criteria of the National Cancer Institute (NCI CTCAE v4).
4. Left ventricular ejection fraction> 39%
5. Adult subjects who have voluntarily signed informed consent before the first study intervention.
6. Minor subjects whose representative / legal guardian has voluntarily signed informed consent before the first study intervention.
7. For mature minors (12 to 17 years old), in addition to the consent signed by the legal guardian, the assent of the child will be obtained.
8. Women of childbearing potential must have a negative pregnancy test at the time inclusion and must agree to use highly effective contraceptive methods (diaphragms plus spermicide or male condom plus spermicide, combined oral contraceptive with a second method of contraceptive implant, injectable contraceptive, permanent intrauterine device, sexual abstinence or partner with vasectomy) while participating in the study and 30 days after the last visit.
9. Presence of a haploidentical donor

Exclusion Criteria:

1. Patients with a history of poor treatment compliance
2. Patients who after a psycho-social assessment are censored as unfit for procedure:

   * Socio-familiar situation that precludes proper participation in the study.
   * Patients with emotional or psychological problems secondary to the illness such as PTSD, phobias, delusions, psychosis, requiring assistance by specialists.
   * Evaluation of the involvement of the family in the patient's health.
   * Inability to understand the information about the trial.
3. Severe (4) organ functional impairment (liver, kidney, respiratory) according to the criteria of the National Cancer Institute (NCI CTCAE v4).
4. They should be considered contraindications, interactions, precautions for use and dose reductions indicated in the respective data sheets.
5. Subjects who have been administered other investigational drugs within 90 days prior to inclusion

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2016-05; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Relapse-free rate after allogeneic haploidentical NK cell infusion | Relapse-free rate at 1 month
  Relapse-free rate according to the clinical guidelines. A bone narrow aspirate one month after NK cell infusion will be evaluated for cytomorphological criteria and minimal residue disease (cytometry or real time PCR). Relapse defined as myeloid blast bone marrow presence with the same diagnosis markers, new ones or mixed. From cytologic analysis 25% of blast or minimal residue disease by cytometry (0,01%) and/or molecular level (0,0001%) present at diagnosis with or without cytogenetic alterations.
Relapse-free rate after allogeneic haploidentical NK cell infusion | Relapse-free rate at one year
  Relapse-free rate according to the clinical guidelines. A bone narrow aspirate one month after NK cell infusion and at least once a year during the three-year follow-up will be evaluated for cytomorphological criteria and minimal residue disease (cytometry or real time PCR). Relapse defined as myeloid blast bone marrow presence with the same diagnosis markers, new ones or mixed. From cytologic analysis 25% of blast or minimal residue disease by cytometry (0,01%) and/or molecular level (0,0001%) present at diagnosis with or without cytogenetic alterations.
Relapse-free rate after allogeneic haploidentical NK cell infusion | Relapse-free rate at two years
  Relapse-free rate according to the clinical guidelines. A bone narrow aspirate one month after NK cell infusion and at least once a year during the three-year follow-up will be evaluated for cytomorphological criteria and minimal residue disease (cytometry or real time PCR). Relapse defined as myeloid blast bone marrow presence with the same diagnosis markers, new ones or mixed. From cytologic analysis 25% of blast or minimal residue disease by cytometry (0,01%) and/or molecular level (0,0001%) present at diagnosis with or without cytogenetic alterations.
Relapse-free rate after allogeneic haploidentical NK cell infusion | Relapse-free rate at three years
  Relapse-free rate according to the clinical guidelines. A bone narrow aspirate one month after NK cell infusion and at least once a year during the three-year follow-up will be evaluated for cytomorphological criteria and minimal residue disease (cytometry or real time PCR). Relapse defined as myeloid blast bone marrow presence with the same diagnosis markers, new ones or mixed. From cytologic analysis 25% of blast or minimal residue disease by cytometry (0,01%) and/or molecular level (0,0001%) present at diagnosis with or without cytogenetic alterations.

SECONDARY OUTCOMES:
Adverse events of special interest: administration issues, infections, immunological/allergic/toxic reactions and concomitant drug interactions. | three years
  All adverse events (AE) will be monitorized. AE of special interest: administration issues, infections, immunological/allergic/toxic reactions and concomitant drug interactions. AE will be classified according to the National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTC) v4.0 criteria or MedDRA classification (mild, moderate, severe or life threatening ).
Evaluation of donor phenotype by SS-PCR | Three years
  Donor HLA phenotype will be determined by SS-PCR. The aim is identify KIR ligand mismatch between donor and recipient to achieve better response. Ideally we will choose KIR ligand mismatch recipient donor pair (http://www.ncbi.nlm.nih.gov/pubmed/26341478).
Evaluation of patient HLA phenotype by SS-PCR | Three years
  Patient HLA phenotype will be determined by SS-PCR. The aim is identify KIR ligand mismatch between donor and recipient to achieve better response. Ideally we will choose KIR ligand mismatch recipient donor pair (http://www.ncbi.nlm.nih.gov/pubmed/26341478).
Evaluation of donor KIR haplotype by PCR | Three years
  The objective is to identify activating KIRs and B haplotype (cen B), by PCR. Ideally we will choose B haplotype donors (http://www.ncbi.nlm.nih.gov/pubmed/20581313)
Analysis of Hematopoietic chimerism after NK infusion by PCR or flow cytometry | Three years
  Chimerism after NK cell infusion by PCR or flow cytometry: to correlate with NK survival and expansion and with clinical outcome (http://www.ncbi.nlm.nih.gov/pubmed/26772158).
Ligand expression of the activatory (MICA, MICB and ULBPs) or inhibitory (HLA-1) receptors of the NK cells | Three years
  Ligand expression of the activatory (MICA, MICB and ULBPs) or inhibitory (HLA-1) receptors of the NK cells will be determined by multiparametric flow cytometry in order to determine the main variables to predict treatment effectiveness and safety.
NK cytotoxic activity | Three years
  In vitro allogenic NK cytotoxic activity against leukemic blast will be performed by real time Eur-TDA fluorescence (Blomberg et al. J Immunol Methods 1986).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pérez Martínez, MD, PhD., Study Chair — aperezmartinez@salud.madrid.org
Locations (6):
- Spain (6):
  - Hospital Universitario de Cruces, Barakaldo, Vizcaya
  - Hospital Materno Infantil de Badajoz, Badajoz
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Materno-Infantil de Málaga, Málaga
  - Hospital de la Arrixaca, Murcia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blomberg K, Granberg C, Hemmila I, Lovgren T. Europium-labelled target cells in an assay of natural killer cell activity. II. A novel non-radioactive method based on time-resolved fluorescence. significance and specificity of the method. J Immunol Methods. 1986 Aug 21;92(1):117-23. doi: 10.1016/0022-1759(86)90511-9. PMID 3745921
- [Derived] Gomez Garcia LM, Escudero A, Mestre C, Fuster Soler JL, Martinez AP, Vagace Valero JM, Vela M, Ruz B, Navarro A, Fernandez L, Fernandez A, Leivas A, Martinez-Lopez J, Ferreras C, De Paz R, Blanquer M, Galan V, Gonzalez B, Corral D, Sisinni L, Mirones I, Balas A, Vicario JL, Valle P, Borobia AM, Perez-Martinez A. Phase 2 Clinical Trial of Infusing Haploidentical K562-mb15-41BBL-Activated and Expanded Natural Killer Cells as Consolidation Therapy for Pediatric Acute Myeloblastic Leukemia. Clin Lymphoma Myeloma Leuk. 2021 May;21(5):328-337.e1. doi: 10.1016/j.clml.2021.01.013. Epub 2021 Jan 25. PMID 33610500
- [Derived] Munoz Builes M, Vela Cuenca M, Fuster Soler JL, Astigarraga I, Pascual Martinez A, Vagace Valero JM, Tong HY, Valentin Quiroga J, Fernandez Casanova L, Escudero Lopez A, Sisinni L, Blanquer M, Mirones Aguilar I, Gonzalez Martinez B, Borobia AM, Perez-Martinez A. Study protocol for a phase II, multicentre, prospective, non-randomised clinical trial to assess the safety and efficacy of infusing allogeneic activated and expanded natural killer cells as consolidation therapy for paediatric acute myeloblastic leukaemia. BMJ Open. 2020 Jan 8;10(1):e029642. doi: 10.1136/bmjopen-2019-029642. PMID 31919123
- See also: Genetics Home Reference — https://ghr.nlm.nih.gov/
- See also: Acute Myeloid Leukemia MedlinePlus — https://www.nlm.nih.gov/medlineplus/acutemyeloidleukemia.html